CLINICAL TRIAL: NCT07233564
Title: Comparison of Pain Between Supraperiosteal Injection of Dexamethasone Versus Placebo on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Comparison of Pain Between Supraperiosteal Injection of Dexamethasone Versus Placebo on Postoperative Pain in Teeth With Symptomatic Irreversible Pulpitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Aqsa Afzal, AAfzal, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 117-ERB/023
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Irreversible Pulpitis
Keywords: Effect of dexamthasone on irreversible pulpitis
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone injection group (Experimental): participant in this arm will receive a supraperiosteal injection of 4mg/ml dexamethasone at the mucobuccal fold prior to endodontic treatment for symptomatic irreversible pulpitis
  Interventions: Drug: Dexamathsone 4mg/ml associated with experimental arm
- Saline injector(placebo) group (Placebo Comparator)
  Interventions: Drug: Normal saline injection

INTERVENTIONS:
Drug: Dexamathsone 4mg/ml associated with experimental arm — particappant in this group will receive a supraperiosteal injection of dexamethasone 4mg/ml at the mucbuccal fold before endodontic treatment of teeth with symptomatic irreversible pulpitis
  Arms: Dexamethasone injection group
Drug: Normal saline injection — particapant in this group will receive a supraperiosteal injection of normal saline at mucobuccal fold in the similar manner and volume as the experoimental drug
  Arms: Saline injector(placebo) group

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of supra periosteal injection of dexamethasone versus placebo in reducing post operative pain in teeth diagnosed with symptomatic irreversible pulpitis. A total of 44 patients will be randomly assigned into two groups: Group A will receive a supra periosteal injection of dexamethasone(4mg/ml), and Group B will receive a similar injection of normal saline as placebo. post operative pain will be assessed at 6hr,24hr and 48hr using a VAS Analogue Scale, with the final outcome measured at 24hrs. the study will help determine whether local dexamethasone injection is effective in minimizing postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or above 18 year old (to have complete apex formation)
* Patient with normal periapical area (no pain on percussion).
* Patient who have not received any preoperative analgesic and antibiotic in last one month.

Exclusion Criteria:

* Pregnancy and Lactation because radiographs are contraindicated.
* Moderate to severe periodontal disease because teeth are not salvageable.
* Patient with nonvital teeth diagnose via cold test and EPT.
* Patient with known sensitivity to dexamethasone by history.
* Patients whose medical history include a history of certain illnesses, such as HIV, heart disease, or epilepsy (conditions that can affect a patient's rate of healing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 24hr after endodontic treatment
  Pain will be measured using a 10 - point Visual Analogue Scale where 0=no pain, 1-3=mild pain, 4-6= moderate pain, and 7-10 = severe pain the absence of pain will be considered as effective treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Saidu College of Dentistry, Swāt, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.1111/j.1875-595X.2011.00092.x